CLINICAL TRIAL: NCT06751485
Title: A Randomized, Open-Label, Parallel-Controlled, Multi-center Phase Ⅲ Study of JSKN003 Versus Investigator-Choice Chemotherapy for Platinum-Resistant, Relapsed Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Brief Title: JSKN003 in Platinum-Resistant, Relapsed Epithelial Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JSKN003-306
Record Dates: First submitted 2024-12-25; First posted 2024-12-30 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Ovarian Cancer; Primary Peritoneal; Fallopian Tube Cancers
Keywords: JSKN003-306
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Doxorubicin; Paclitaxel; Topotecan

STUDY DESIGN:
Intervention Model Description: To evaluate the efficacy and safety of JSKN003 compared with investigator-chosen chemotherapy in patients with platinum-resistant recurrent epithelial ovarian cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Treatment group 1:JSKN003 (Experimental): Drug: JSKN003 JSKN003 dose 1
  Interventions: Drug: JSKN003
- Active Comparator: Treatment group 2: Investigator's choice of chemotherapy (Active Comparator): Drug: Doxorubicin Doxorubicin dose 2
  Drug: Paclitaxel Paclitaxel dose 3
  Drug: Topotecan Topotecan dose 4
  Interventions: Drug: Doxorubicin; Drug: Paclitaxel; Drug: Topotecan

INTERVENTIONS:
Drug: JSKN003 — Experimental drug
  Arms: Experimental: Treatment group 1:JSKN003
Drug: Doxorubicin — Active Comparator
  Arms: Active Comparator: Treatment group 2: Investigator's choice of chemotherapy
Drug: Paclitaxel — Active Comparator
  Arms: Active Comparator: Treatment group 2: Investigator's choice of chemotherapy
Drug: Topotecan — Active Comparator
  Arms: Active Comparator: Treatment group 2: Investigator's choice of chemotherapy

SUMMARY:
This study is a randomized, open-label, controlled, phase III study to evaluate the efficacy and safety of JSKN003 versus investigator's choice of chemotherapy in patients with platinum-resistant, relapsed epithelial Ovarian, primary peritoneal, or fallopian tube cancer.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation and written informed consent.
* ≥18 years;
* Histologically confirmed epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.
* Confirmed platinum-resistant relapse.
* According to RECIST 1.1 criteria, there must be at least one measurable lesion in the baseline.
* Expected survival of more than 3 months.
* ECOG performance status score of 0 or 1.
* Adequate organ function.
* Capable and willing to comply with the study protocol, treatment plan, laboratory tests, and other related study procedures.

Exclusion Criteria:

* Primary platinum-refractory disease.
* Active central nervous system metastases.
* Uncontrolled pleural effusion.
* Previous treatment with topoisomerase I inhibitor ADCs.
* Other malignant tumors within 5 years.
* Interstitial pneumonia/lung disease requiring systemic corticosteroids or suspected interstitial pneumonia/lung disease.
* Uncontrolled comorbidities.
* Toxicity from previous anti-cancer treatments not recovered to CTCAE Grade ≤1.
* History of allogeneic bone marrow or organ transplantation.
* Allergic reactions or hypersensitivity to antibody drugs.
* Conditions affecting study drug treatment safety or compliance, including psychiatric disorders, alcohol abuse, or drug abuse.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) assessed by Blinded Independent Review Committee (BIRC) as per RECIST 1.1 | Up to approximately 22 months
  PFS was defined as the time from randomization until the date of progressive disease or death, whichever occurred first

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 22 months
  OS was defined as the time from the date of first dose until the date of death from any cause
Overall Response Rate (ORR) evaluated by BIRC as per RECIST 1.1 | Up to approximately 22 months
  ORR was defined as the proportion of subjects achieving Complete Response (CR) or Partial Response (PR)
Duration of Response (DoR) evaluated by BIRC as per RECIST 1.1 | Up to approximately 22 months
  DOR was defined as the time from CR/PR to PD or death from any cause, whichever occurs first
Disease Control Rate (DCR) evaluated by BIRC as per RECIST 1.1 | Up to approximately 22 months
  DCR was defined as the proportion of subjects whose best overall response is CR, PR, or Stable Disease (SD)
PFS evaluated by the Investigator as per RECIST 1.1 | Up to approximately 22 months
  PFS was defined as the time from randomization until the date of progressive disease or death, whichever occurred first
ORR evaluated by the Investigator as per RECIST 1.1 | Up to approximately 22 months
  ORR was defined as the proportion of subjects achieving Complete Response (CR) or Partial Response (PR)
DoR evaluated by the Investigator as per RECIST 1.1 | Up to approximately 22 months
  DOR was defined as the time from CR/PR to PD or death from any cause, whichever occurs first
DCR evaluated by the Investigator as per RECIST 1.1 | Up to approximately 22 months
  DCR was defined as the proportion of subjects whose best overall response is CR, PR, or Stable Disease (SD)
CA-125 Response Rate assessed by the Gynaecologic Cancer Intergroup (GCIG) criteria | Up to approximately 22 months
  CA-125 Response Rate was assessed according to the GCIG criteria
Number and Severity of Treatment-emergent Adverse Events (TEAEs) | Up to approximately 22 months
  The incidence and severity of TEAEs and TRAEs (Treatment-related Adverse Events, graded according to NCI CTCAE 5.0), Serious AEs (SAEs), laboratory tests, etc.

IPD SHARING:
Plan to Share IPD: Undecided